CLINICAL TRIAL: NCT06183372
Title: A Randomised Double-blind Placebo-controlled Acute Trial of Encapsulated Lemon Balm Efficacy and Tolerance on Calmness and Mood During Periods of Cognitive Demand
Brief Title: Enhancement of Calmness and Mood Following Acute Lemon Balm Supplementation During Cognitive Demand in Adults
Acronym: LemCog
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Naturex (Other)
Responsible Party: Principal Investigator, Prof Claire Williams, Chair of Neuroscience, University of Reading
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 23/25
Record Dates: First submitted 2023-12-13; First posted 2023-12-27 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Stress; Mood Disturbance
Keywords: Calmness; Subject Satisfaction; Mood enhancement; Relaxation; Lemon Balm; Melissa Officinalis; Herbal Psychotropic; Cognitive demand; Memory; Attention; Executive Function
MeSH Terms: interventions — lemon balm leaf extract

STUDY DESIGN:
Intervention Model Description: Between- and within-groups (mixed) model
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lemon balm (Experimental): 300mg Lemon balm and Maltoxdextrin capsules
  Interventions: Dietary Supplement: Lemon balm
- Placebo (Placebo Comparator): 300mg Maltodextrin capsules
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Lemon balm — 300mg Lemon balm and Maltoxdextrin capsules Other Name: Melissa Officinalis L.
  Arms: Lemon balm
Dietary Supplement: Placebo — 300mg Maltodextrin capsules
  Arms: Placebo

SUMMARY:
This study aims to investigate the effect of a single dose (300mg) of encapsulated aqueous lemon balm extract on measures of calmness and mood during periods of cognitive demand over the course of the day in healthy adults aged 18-40 years with moderate stress (PSS entry between 14 to 26).

DETAILED DESCRIPTION:
Cognitive overload can be a common occurrence in an information saturated world (Eppler et al., 2008; Graf et al., 2021; Pass et al., 2004), and chronic cognitive overload is considered an initiating step in the emergence of various physical and emotional health concerns, likely due to high processing demands on the working memory neural system (Graf et al., 2021). Over time, psychological and physiological stress may arise, however current chemical interventions may be unsuitable for those experiencing mild-to-moderate levels of stress (Ghazizadeh et al., 2021). Indeed, long-term use of psychotropic medicines have previously been associated with a worsening of psychological symptoms (Bertuccioli et al., 2022). Therefore, identifying interventions for those experiencing mild-to-moderate stress will have strong public health implications for the prevention or reduction of symptoms. In addition, an opportunity for dietary supplementation as an over-the-counter option for those who do not wish to take chemical interventions is becoming a popular choice (Ghazizadeh et al., 2021; Bertuccioli et al. 2022).

The current study will employ a parallel, double-blind, randomised placebo-controlled trial, assessing the effect of a single dose intervention of lemon balm extract (or matched placebo) in young-to-middle-aged adults with moderate levels of perceived stress. Subjects will be pre-screened to determine eligibility using the perceived stress questionnaire, where scores between 14 to 26 are indicative of moderate stress, to provide a total of 130 participants. The study comprises a familiarisation visit followed by an acute test day at the Nutritional Psychology Unit based at the University of Reading. The familiarisation visit will allow participants to practice the cognitive battery, complete calmness and mood measures, and provide information on habitual diet (Epic-Norfolk FFQ) and general health and lifestyle patterns to confirm eligibility. On the acute test day, subjective calmness and mood ratings will be recorded at various timepoints throughout the day, beginning with an initial baseline measurement (0h), and then 1h, 3h and 5h after consuming an acute dose of lemon balm extract (300mg) or a matched placebo. At these same timepoints, a computer-based cognitive battery will be completed, consisting of several tasks assessing domains of executive function, attention and memory. On the acute test day participants will arrive fasted and will be provided with a standardised breakfast (two croissants and a glass of water) to be consumed prior to 0h baseline measures. A standardised lunch (cheese sandwich, packet of crisps, and water) will also be provided after the 3h timepoint.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, between 18-40 years old
* Moderate Stress problems (PSS between 14 to 26)
* No alcohol or vigorous activity 24h before the task
* No coffee/caffeine intake 12h before the visits
* Non-smokers or Must not smoke during 7 days prior to the trial: Includes smoking tobacco, vaping nicotine, using nicotine replacement products, or occasional social smoking.
* Willingness to wash out for food supplementation during 2 weeks before the experiment

Exclusion Criteria:

* Use medications that may affect the outcome
* Any long-term psychological or physiological health conditions
* Have any allergic reactions to ingredients in the capsules
* Have a BMI greater than or equal to 30
* Have any allergic reactions to ingredients in the capsules
* Consumed more than 400 mg of caffeine (>5 expresso) per day in the past 2 weeks
* Have used any psychotropic medications, stimulants, cannabis, non-registered drug products, or illicit substances in the past 2 weeks, were at risk of drug or alcohol abuse
* Taking any dietary supplements which they are unwilling to stop for the duration of the study
* Have sleep disorders or are taking sleep aid medication
* Fail to demonstrate adequate minimal performance on lab, computer-based cognitive tasks
* Have a diagnosed neurological condition, or learning/behavioural or neurodevelopmental differences (e.g. dyslexia, autism, ADHD).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2023-12-02 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Calmness 9-point Likert Scale | Baseline
  A validated 9-point Likert scale with Calmness Anchor points (CAP) ranging from 1, "Not at all Calm" to 9, "Extremely Calm"
Calmness 9-point Likert Scale | 5 hours following intervention
  A validated 9-point Likert scale with Calmness Anchor points (CAP) ranging from 1, "Not at all Calm" to 9, "Extremely Calm"

SECONDARY OUTCOMES:
Fatigue 9-point Likert Scale | Baseline
  A validated 9-point Likert scale with Fatigue Anchor points (FAP) ranging from 1, "Not at all mentally fatigued" and 9, "Extremely mentally fatigued"
Fatigue 9-point Likert Scale | 5 hours following intervention
  A validated 9-point Likert scale with Fatigue Anchor points (FAP) ranging from 1, "Not at all mentally fatigued" and 9, "Extremely mentally fatigued"
Subject Satisfaction 4-point Category Scale | 1 hour following intervention
  A two-part questionnaire based on a previously published 4-category rating questionnaire. The first part asks about current levels of tiredness and mental overload, using a 4-point Likert anchored from "not at all" (score 1) to "extremely" (score 4). The second part asks how satisfied a person is with their levels of tiredness and mental overload following supplementation, and asks them to rate their overall satisfaction with the supplement, using scales "not at all satisfied" (score 1) to "entirely satisfied" (score 4).
Subject Satisfaction 4-point Category Scale | 3 hours following intervention
  A two-part questionnaire based on a previously published 4-category rating questionnaire. The first part asks about current levels of tiredness and mental overload, using a 4-point Likert anchored from "not at all" (score 1) to "extremely" (score 4). The second part asks how satisfied a person is with their levels of tiredness and mental overload following supplementation, and asks them to rate their overall satisfaction with the supplement, using scales "not at all satisfied" (score 1) to "entirely satisfied" (score 4).
Subject Satisfaction 4-point Category Scale | 5 hours following intervention
  A two-part questionnaire based on a previously published 4-category rating questionnaire. The first part asks about current levels of tiredness and mental overload, using a 4-point Likert anchored from "not at all" (score 1) to "extremely" (score 4). The second part asks how satisfied a person is with their levels of tiredness and mental overload following supplementation, and asks them to rate their overall satisfaction with the supplement, using scales "not at all satisfied" (score 1) to "entirely satisfied" (score 4).
Visual Analogue Stress Scale | Baseline
  Ratings of stress are captured using 100mm Visual Analogue Scales anchored at each end by words descriptive of the minimal and maximal extremes of one statement (unipolar). On this linear scale, the person indicates how he or she is feeling at the moment by placing a mark between 2 statements concerning a specific condition of the dimension being measured. This brief instrument assesses levels of stress, anxiety, calmness and relaxation. Individual scores are combined to form 'stress/anxiety' and 'calm/relaxed' scores, where a higher score (average % along the line) represents more of the respective descriptor.
Visual Analogue Stress Scale | 1 hour following intervention
  Ratings of stress are captured using 100mm Visual Analogue Scales anchored at each end by words descriptive of the minimal and maximal extremes of one statement (unipolar). On this linear scale, the person indicates how he or she is feeling at the moment by placing a mark between 2 statements concerning a specific condition of the dimension being measured. This brief instrument assesses levels of stress, anxiety, calmness and relaxation. Individual scores are combined to form 'stress/anxiety' and 'calm/relaxed' scores, where a higher score (average % along the line) represents more of the respective descriptor.
Visual Analogue Stress Scale | 3 hours following intervention
  Ratings of stress are captured using 100mm Visual Analogue Scales anchored at each end by words descriptive of the minimal and maximal extremes of one statement (unipolar). On this linear scale, the person indicates how he or she is feeling at the moment by placing a mark between 2 statements concerning a specific condition of the dimension being measured. This brief instrument assesses levels of stress, anxiety, calmness and relaxation. Individual scores are combined to form 'stress/anxiety' and 'calm/relaxed' scores, where a higher score (average % along the line) represents more of the respective descriptor.
Visual Analogue Stress Scale | 5 hours following intervention
  Ratings of stress are captured using 100mm Visual Analogue Scales anchored at each end by words descriptive of the minimal and maximal extremes of one statement (unipolar). On this linear scale, the person indicates how he or she is feeling at the moment by placing a mark between 2 statements concerning a specific condition of the dimension being measured. This brief instrument assesses levels of stress, anxiety, calmness and relaxation. Individual scores are combined to form 'stress/anxiety' and 'calm/relaxed' scores, where a higher score (average % along the line) represents more of the respective descriptor.
Bond-Lader 16-item Visual Analogue Stress Scale | Baseline
  A widely used 16-item tool for measuring transient mood where 100mm scales anchored by various antonyms (e.g. Alert-Drowsy, Lethargic-Energetic) and are then clustered into respective mood factors alertness, calmness and contentedness
Bond-Lader 16-item Visual Analogue Stress Scale | 1 hour following intervention
  A widely used 16-item tool for measuring transient mood where 100mm scales anchored by various antonyms (e.g. Alert-Drowsy, Lethargic-Energetic) and are then clustered into respective mood factors alertness, calmness and contentedness
Bond-Lader 16-item Visual Analogue Stress Scale | 3 hours following intervention
  A widely used 16-item tool for measuring transient mood where 100mm scales anchored by various antonyms (e.g. Alert-Drowsy, Lethargic-Energetic) and are then clustered into respective mood factors alertness, calmness and contentedness
Bond-Lader 16-item Visual Analogue Stress Scale | 5 hours following intervention
  A widely used 16-item tool for measuring transient mood where 100mm scales anchored by various antonyms (e.g. Alert-Drowsy, Lethargic-Energetic) and are then clustered into respective mood factors alertness, calmness and contentedness
Immediate Word Recall (Rey Auditory Verbal Learning Task) | Baseline
  A standardised cognitive measure to episodic memory. In this task participants are visually presented with a sequential list of fifteen words where they are then given 1 minute to type as many words as they can remember. At each sitting of the task, a different word list will be presented which will be matched for linguistic familiarity, concreteness and frequency. The dependent variable is the number of words correctly recalled.
Immediate Word Recall (Rey Auditory Verbal Learning Task) | 1 hour following intervention
  A standardised cognitive measure to episodic memory. In this task participants are visually presented with a sequential list of fifteen words where they are then given 1 minute to type as many words as they can remember. At each sitting of the task, a different word list will be presented which will be matched for linguistic familiarity, concreteness and frequency. The dependent variable is the number of words correctly recalled.
Immediate Word Recall (Rey Auditory Verbal Learning Task) | 3 hours following intervention
  A standardised cognitive measure to episodic memory. In this task participants are visually presented with a sequential list of fifteen words where they are then given 1 minute to type as many words as they can remember. At each sitting of the task, a different word list will be presented which will be matched for linguistic familiarity, concreteness and frequency. The dependent variable is the number of words correctly recalled.
Immediate Word Recall (Rey Auditory Verbal Learning Task) | 5 hours following intervention
  A standardised cognitive measure to episodic memory. In this task participants are visually presented with a sequential list of fifteen words where they are then given 1 minute to type as many words as they can remember. At each sitting of the task, a different word list will be presented which will be matched for linguistic familiarity, concreteness and frequency. The dependent variable is the number of words correctly recalled.
Delayed Word Recall (Rey Auditory Verbal Learning Task) | Baseline
  A standardised cognitive measure to assess the level of delayed episodic memory. Participants will be required to type as many words as they can remember from the immediate word recall presentation after a delay of approximately 30 minutes following the initial presentation. The dependent variable is the number of words correctly recalled.
Delayed Word Recall (Rey Auditory Verbal Learning Task) | 1 hour following intervention
  A standardised cognitive measure to assess the level of delayed episodic memory. Participants will be required to type as many words as they can remember from the immediate word recall presentation after a delay of approximately 30 minutes following the initial presentation. The dependent variable is the number of words correctly recalled.
Delayed Word Recall (Rey Auditory Verbal Learning Task) | 3 hours following intervention
  A standardised cognitive measure to assess the level of delayed episodic memory. Participants will be required to type as many words as they can remember from the immediate word recall presentation after a delay of approximately 30 minutes following the initial presentation. The dependent variable is the number of words correctly recalled.
Delayed Word Recall (Rey Auditory Verbal Learning Task) | 5 hours following intervention
  A standardised cognitive measure to assess the level of delayed episodic memory. Participants will be required to type as many words as they can remember from the immediate word recall presentation after a delay of approximately 30 minutes following the initial presentation. The dependent variable is the number of words correctly recalled.
Modified Attention Network Task (with two blocks of Serial 3's) | Baseline
  A standardised measure to assess executive function and attention. In this task participants respond to the direction of a centrally presented arrow by pressing the corresponding left and right arrow keys. Across multiple trials, the target stimuli are either flanked by arrows pointing in the same direction (congruent) or opposite (incongruent). The number of flanking arrows also varies between trials (load). Two blocks are presented. In the second block, participants will be distracted by noise through headphones. In addition, during further subsections of the ANT an oral serial 3 (S3) subtractions task will also be performed to further assess attention and working memory function. In this S3 task participants subtract backwards starting with the number 50 until they can go no further. The S3 performance will be in place to add additional cognitive load and the dependent variable will be ANT performance (accuracy and reaction time) under varying conditions of congruency and load.
Modified Attention Network Task (with two blocks of Serial 3's) | 1 hour following intervention
  A standardised measure to assess executive function and attention. In this task participants respond to the direction of a centrally presented arrow by pressing the corresponding left and right arrow keys. Across multiple trials, the target stimuli are either flanked by arrows pointing in the same direction (congruent) or opposite (incongruent). The number of flanking arrows also varies between trials (load). Two blocks are presented. In the second block, participants will be distracted by noise through headphones. In addition, during further subsections of the ANT an oral serial 3 (S3) subtractions task will also be performed to further assess attention and working memory function. In this S3 task participants subtract backwards starting with the number 50 until they can go no further. The S3 performance will be in place to add additional cognitive load and the dependent variable will be ANT performance (accuracy and reaction time) under varying conditions of congruency and load.
Modified Attention Network Task (with two blocks of Serial 3's) | 3 hours following intervention
  A standardised measure to assess executive function and attention. In this task participants respond to the direction of a centrally presented arrow by pressing the corresponding left and right arrow keys. Across multiple trials, the target stimuli are either flanked by arrows pointing in the same direction (congruent) or opposite (incongruent). The number of flanking arrows also varies between trials (load). Two blocks are presented. In the second block, participants will be distracted by noise through headphones. In addition, during further subsections of the ANT an oral serial 3 (S3) subtractions task will also be performed to further assess attention and working memory function. In this S3 task participants subtract backwards starting with the number 50 until they can go no further. The S3 performance will be in place to add additional cognitive load and the dependent variable will be ANT performance (accuracy and reaction time) under varying conditions of congruency and load.
Modified Attention Network Task (with two blocks of Serial 3's) | 5 hours following intervention
  A standardised measure to assess executive function and attention. In this task participants respond to the direction of a centrally presented arrow by pressing the corresponding left and right arrow keys. Across multiple trials, the target stimuli are either flanked by arrows pointing in the same direction (congruent) or opposite (incongruent). The number of flanking arrows also varies between trials (load). Two blocks are presented. In the second block, participants will be distracted by noise through headphones. In addition, during further subsections of the ANT an oral serial 3 (S3) subtractions task will also be performed to further assess attention and working memory function. In this S3 task participants subtract backwards starting with the number 50 until they can go no further. The S3 performance will be in place to add additional cognitive load and the dependent variable will be ANT performance (accuracy and reaction time) under varying conditions of congruency and load.
Task Switching Test | Baseline
  A standardised cognitive task to assess executive function. In this task participants are presented with a computerised visual circle with 8 equally spaced radii that form 8 segments, 4 above and 4 below a bold line. A stimulus digit appears sequentially in each segment in a clockwise direction. If the digit was located above the bold line, participants then indicate whether the digit was odd or even using labelled arrow keys (left for odd, right for even). When the digit is below the bold line, participants again use the arrow keys to indicate whether the digit is higher or lower than 5 (left for higher, right for lower). The dependent variable will be TST performance (accuracy and reaction time) across all trials, and comparing switch trials (where the rule changes from the previous trial) and non-switch trials (where the rule stays the same as the previous trial).
Task Switching Test | 1 hours following intervention
  A standardised cognitive task to assess executive function. In this task participants are presented with a computerised visual circle with 8 equally spaced radii that form 8 segments, 4 above and 4 below a bold line. A stimulus digit appears sequentially in each segment in a clockwise direction. If the digit was located above the bold line, participants then indicate whether the digit was odd or even using labelled arrow keys (left for odd, right for even). When the digit is below the bold line, participants again use the arrow keys to indicate whether the digit is higher or lower than 5 (left for higher, right for lower). The dependent variable will be TST performance (accuracy and reaction time) across all trials, and comparing switch trials (where the rule changes from the previous trial) and non-switch trials (where the rule stays the same as the previous trial).
Task Switching Test | 3 hours following intervention
  A standardised cognitive task to assess executive function. In this task participants are presented with a computerised visual circle with 8 equally spaced radii that form 8 segments, 4 above and 4 below a bold line. A stimulus digit appears sequentially in each segment in a clockwise direction. If the digit was located above the bold line, participants then indicate whether the digit was odd or even using labelled arrow keys (left for odd, right for even). When the digit is below the bold line, participants again use the arrow keys to indicate whether the digit is higher or lower than 5 (left for higher, right for lower).The dependent variable will be TST performance (accuracy and reaction time) across all trials, and comparing switch trials (where the rule changes from the previous trial) and non-switch trials (where the rule stays the same as the previous trial).
Task Switching Test | 5 hours following intervention
  A standardised cognitive task to assess executive function. In this task participants are presented with a computerised visual circle with 8 equally spaced radii that form 8 segments, 4 above and 4 below a bold line. A stimulus digit appears sequentially in each segment in a clockwise direction. If the digit was located above the bold line, participants then indicate whether the digit was odd or even using labelled arrow keys (left for odd, right for even). When the digit is below the bold line, participants again use the arrow keys to indicate whether the digit is higher or lower than 5 (left for higher, right for lower).The dependent variable will be TST performance (accuracy and reaction time) across all trials, and comparing switch trials (where the rule changes from the previous trial) and non-switch trials (where the rule stays the same as the previous trial).
Rapid Visual Information Processing Task | Baseline
  A standardised cognitive task which involves presenting a series of digits on screen in quick succession. The participant will then be required to monitor the digits for sequences of three consecutive even or three consecutive odd digits. To indicate the end of a target sequence, participants will press the space bar as quickly as possible. The dependent variable is task performance (accuracy and reaction time).
Rapid Visual Information Processing Task | 1 hour following intervention
  A standardised cognitive task which involves presenting a series of digits on screen in quick succession. The participant will then be required to monitor the digits for sequences of three consecutive even or three consecutive odd digits. To indicate the end of a target sequence, participants will press the space bar as quickly as possible. The dependent variable is task performance (accuracy and reaction time).
Rapid Visual Information Processing Task | 3 hours following intervention
  A standardised cognitive task which involves presenting a series of digits on a screen in quick succession. The participant will then be required to monitor the digits for sequences of three consecutive even or three consecutive odd digits. To indicate the end of a target sequence, participants will press the space bar as quickly as possible. The dependent variable is task performance (accuracy and reaction time).
Rapid Visual Information Processing Task | 5 hours following intervention
  A standardised cognitive task which involves presenting a series of digits on a screen in quick succession. The participant will then be required to monitor the digits for sequences of three consecutive even or three consecutive odd digits. To indicate the end of a target sequence, participants will press the space bar as quickly as possible. The dependent variable is task performance (accuracy and reaction time).
Paced Auditory Serial Addition Task | Baseline
  A standardised cognitive task to assess attention and memory. The participant is presented with a string of auditory single digits and required to add each new digit to the one immediately prior to it out loud so that responses can be recorded. The dependent variable is therefore accuracy of calculation. The task comprises of 4, 2 minute blocks, where interstimulus time progressively decreases from 2.8 seconds to 1.6 seconds and cognitive demand therefore progressively increases.
Paced Auditory Serial Addition Task | 1 hour following intervention
  A standardised cognitive task to assess attention and memory. The participant is presented with a string of auditory single digits and required to add each new digit to the one immediately prior to it out loud so that responses can be recorded. The dependent variable is therefore accuracy of calculation. The task comprises of 4, 2 minute blocks, where interstimulus time progressively decreases from 2.8 seconds to 1.6 seconds and cognitive demand therefore progressively increases.
Paced Auditory Serial Addition Task | 3 hours following intervention
  A standardised cognitive task to assess attention and memory. The participant is presented with a string of auditory single digits and required to add each new digit to the one immediately prior to it out loud so that responses can be recorded. The dependent variable is therefore accuracy of calculation. The task comprises of 4, 2 minute blocks, where interstimulus time progressively decreases from 2.8 seconds to 1.6 seconds and cognitive demand therefore progressively increases.
Paced Auditory Serial Addition Task | 5 hours following intervention
  A standardised cognitive task to assess attention and memory. The participant is presented with a string of auditory single digits and required to add each new digit to the one immediately prior to it out loud so that responses can be recorded. The dependent variable is therefore accuracy of calculation. The task comprises of 4, 2 minute blocks, where interstimulus time progressively decreases from 2.8 seconds to 1.6 seconds and cognitive demand therefore progressively increases.
Systolic Blood Pressure | Baseline
  Average (triplicate) resting brachial left arm cuffed systolic blood pressure mmHg
Systolic Blood Pressure | 1 hour following intervention
  Average (triplicate) resting brachial left arm cuffed systolic blood pressure mmHg
Systolic Blood Pressure | 3 hour following intervention
  Average (triplicate) resting brachial (left arm) cuffed systolic blood pressure mmHg
Systolic Blood Pressure | 5 hour following intervention
  Average (triplicate) resting brachial (left arm) cuffed systolic blood pressure mmHg
Diastolic Blood Pressure | Baseline
  Average (triplicate) resting brachial (left arm) cuffed diastolic blood pressure mmHg
Diastolic Blood Pressure | 1 hour following intervention
  Average (triplicate) resting brachial (left arm) cuffed diastolic blood pressure mmHg
Diastolic Blood Pressure | 3 hours following intervention
  Average (triplicate) resting brachial (left arm) cuffed diastolic blood pressure mmHg
Diastolic Blood Pressure | 5 hours following intervention
  Average (triplicate) resting brachial (left arm) cuffed diastolic blood pressure mmHg
Heart Rate | Baseline
  Average (triplicate) resting brachial (left arm) cuffed heart rate bpm
Heart Rate | 1 hour following intervention
  Average (triplicate) resting brachial (left arm) cuffed heart rate bpm
Heart Rate | 3 hours following intervention
  Average (triplicate) resting brachial (left arm) cuffed heart rate bpm
Heart Rate | 5 hours following intervention
  Average (triplicate) resting brachial (left arm) cuffed heart rate bpm

CONTACTS AND LOCATIONS:
Overall Officials: Claire M Williams, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data may be made available on a platform such as Open Science Framework (www.osf.io) or a data repository linked to academic journals, in accordance with Open Science principles.
Supporting Information: Study Protocol, SAP

REFERENCES:
- [Background] Bertuccioli A, Cardinali M, Di Pierro F, Magi S, Zonzini G. A Practical Perspective on the Use of Botanicals During the COVID-19 Pandemic: From Proven to Potential Interactions. J Med Food. 2022 Jan;25(1):1-11. doi: 10.1089/jmf.2021.0062. Epub 2021 Nov 17. PMID 34788575
- [Background] Ghazizadeh J, Sadigh-Eteghad S, Marx W, Fakhari A, Hamedeyazdan S, Torbati M, Taheri-Tarighi S, Araj-Khodaei M, Mirghafourvand M. The effects of lemon balm (Melissa officinalis L.) on depression and anxiety in clinical trials: A systematic review and meta-analysis. Phytother Res. 2021 Dec;35(12):6690-6705. doi: 10.1002/ptr.7252. Epub 2021 Aug 27. PMID 34449930
- See also: Eppler, M.J., Mengis, J. (2008). The Concept of Information Overload - A Review of Literature from Organization Science... (2004). In: Meckel, M., Schmid, B.F. (eds) Kommunikationsmanagement im Wandel. Gab — https://link.springer.com/chapter/10.1007/978-3-8349-9772-2_15

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-30): https://cdn.clinicaltrials.gov/large-docs/72/NCT06183372/Prot_SAP_000.pdf